CLINICAL TRIAL: NCT07178093
Title: Effects of Antrodia Cinnamomea on the Hepatoma Patients After Transcatheter Hepatic Artery Chemoembolization
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Tzu Chi Hospital (Other)
Responsible Party: Principal Investigator, Yu, Cheng-Chan, Principal Investigator, Taichung Tzu Chi Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REC111-54
Record Dates: First submitted 2023-04-28; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Hepatocellular Carcinoma; Transarterial Chemoembolization
Keywords: hepatocellular carcinoma (HCC), viral hepatitis, Antrodia cinnamomea, post-TACE syndrome; hepatocellular carcinoma; antrodia cinnamomea; post-TACE syndrome
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: Randomized double blind placebo controlled study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antrodia cinnamomea group (Experimental): This group will use Antrodia cinnamomea on the hepatoma patients after Transcatheter hepatic artery chemoembolization. The choice of chemical drug dosage for the patient's hepatic artery embolization is evaluated according to the size of the tumor, which can be divided into 1. Epirubicin 10mg + Lipiodol 10ml 2. Epirubicin 20mg + Lipiodol 10ml; oral dosage form of Antrodia cinnamomea is single capsule/500mg, each oral dose is 2 capsules/1000mg. The experiment lasted for 11 days, and patients were required to take Kangjian Antrodia cinnamomea 3 days before embolization, the day of embolization to the 7th day after surgery, once a day in the morning and evening after meals, 2 capsules each time.
  Interventions: Dietary Supplement: Antrodia cinnamomea
- Placebo group (Placebo Comparator): This group will use placebo on the hepatoma patients after Transcatheter hepatic artery chemoembolization. The choice of chemical drug dosage for the patient's hepatic artery embolization is evaluated according to the size of the tumor, which can be divided into 1. Epirubicin 10mg + Lipiodol 10ml 2. Epirubicin 20mg + Lipiodol 10ml; oral dosage of placebo is 2 capsules twice daily. The experiment lasted for 11 days, and patients were required to take placebo 3 days before embolization, the day of embolization to the 7th day after surgery, once a day in the morning and evening after meals, 2 capsules each time.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Antrodia cinnamomea — The experiment lasted for 11 days, and patients were required to take Kangjian Antrodia cinnamomea 3 days before embolization, the day of embolization to the 7th day after surgery, once a day in the morning and evening after meals, 2 capsules each time.
  Other Names: Antrodia cinnamomea group
  Arms: Antrodia cinnamomea group
Dietary Supplement: placebo — The experiment lasted for 11 days, and patients were required to take placebo 3 days before embolization, the day of embolization to the 7th day after surgery, once a day in the morning and evening after meals, 2 capsules each time.
  Arms: Placebo group

SUMMARY:
Effects of Antrodia cinnamomea on the hepatoma patients after Transcatheter hepatic artery chemoembolization

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) accounts for 7% of all cancers worldwide and is the most common, primary liver malignancy globally. It is the second leading cause of cancer-related mortality in Taiwan. Most of the patients with HCCs are associated with hepatitis virus B or C infection, and combined with abnormal liver function or liver cirrhosis. The treatment of HCC includes curative treatment, including surgical resection, liver transplantation, and radiofrequency ablation. Non-curative treatment includes Transcatheter hepatic artery chemoembolization or medical therapy, such as target therapies or immunotherapies. Some patients suffered from post-TACE syndrome, e.g., abdominal pain, nausea, fever, or impaired liver function, after TACE. The clinical application was limited by the possibility of liver function deterioration. There is no standard treatment for the post-TACE syndrome currently. Therapies capable of liver protection could enhance the safety and effect of TACE.

Antrodia cinnamomea (AC) is a medicinal fungal species that has been widely used as a healthy food in Taiwan for the treatment of diverse health-related conditions, in recognition of its anticancer, hepatoprotective, anti-inflammatory, antidiabetic and neuroprotective activities. The properties of antitumor and hepatoprotective make A. cinnamomea extract or its major compounds an ideal candidate for enhancing the treatment effect for HCC.

Many cancer patients in Taiwan took Antrodia cinnamomea products during the course of therapies. In this study, we want to elucidate the effect of Antrodia cinnamomea on the hepatoma patients after Transcatheter hepatic artery chemoembolization, such as the improvement of post-TACE syndrome ( liver function impairment, fever, nausea, and abdominal pain), the quality of life, and hospital stay, etc.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form
* Aged between 20 and 80
* Child-Pugh score class A, B
* Serum bilirubin level ≤ 1.5 times the upper limit of normal, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels ≤ 2 times the upper limit of normal

Exclusion Criteria:

* Unwillingness to sign the informed consent form
* Child-Pugh score class C
* Patients with main portal vein thrombosis
* Patients with diffuse liver tumors
* Those who are allergic to the contrast medium
* Those with abnormal coagulation function
* Those with severe dysfunction of brain, heart and lung
* Patients with severe renal dysfunction (except those receiving renal dialysis)
* Unable to cooperate
* Those with uncontrolled arrhythmia and unstable blood pressure
* Some patients with abnormal thyroid function
* Any other contraindications such as active gastrointestinal bleeding, refractory ascites, or severe portal hypertension
* Pregnant or lactating women

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of serum Aspartate Transaminase (AST) level after TACE | 28 days
  The serum Aspartate Transaminase (AST) levels after TACE day 1, day 3, day 7, day 28 are compared to the baseline.
Changes of serum Alanine Aminotransferase (ALT) level after TACE | 28 days
  The serum Alanine Aminotransferase (ALT) levels after TACE day 1, day 3, day 7, day 28 are compared to the baseline.
Changes of serum total bilirubin level after TACE | 28 days
  The serum total bilirubin levels after TACE day 1, day 3, day 7, and day 28 are compared to the baseline
Changes of serum albumin level after TACE | 28 days
  The serum albumin levels after TACE day 1, day 3, day 7, and day 28 are compared to the baseline
Changes of prothrombin time after TACE | 28 days
  The prothrombin time after TACE day 1, day 3, day 7, and day 28 are compared to the baseline.

SECONDARY OUTCOMES:
Improvement of the quality of life | 28 days
  European Organisation for Research and Treatment of Cancer Core Quality of Life questionnaire (EORTC QLQ-C30 questionnaire) has 30 items, covering both general health status and cancer-related symptoms. Each item is scored on a 4-point Likert scale (1 = "Not at all" to 4 = "Very much"), except for the global health/QoL items, which use a 7-point scale (1 = "Very poor" to 7 = "Excellent"). The differences of the scores after TACE are recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Tzu-Chi Hospital, Taichung, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No